CLINICAL TRIAL: NCT02952417
Title: Sex Differences in Relative Survival and Excess Mortality Following Acute Myocardial Infarction: National Cohort Study Using the SWEDEHEART Registry
Brief Title: Sex Differences in Relative Survival and Excess Mortality Following Acute Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Oras Alabas, Doctor, University of Leeds
Other Study IDs: 1.001
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — Mortality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- STEMI and NSTEMI Women: Women with ST-segment elevation myocardial infarction (STEMI) and women non-STEMI (NSTEMI) who survived following acute myocardial infarction and at risk of excess mortality.
  Interventions: Other: Excess mortality
- STEMI and NSTEMI Men: Men with ST-segment elevation myocardial infarction (STEMI) and women non-STEMI (NSTEMI) who survived following acute myocardial infarction and at risk of excess mortality.

INTERVENTIONS:
Other: Excess mortality — Relative survival was defined as the observed survival among patients with STEMI and NSTEMI divided by the expected survival in the age, sex and year matched populace of Sweden.
  Groups: STEMI and NSTEMI Women

SUMMARY:
The aim of this study was to estimate the impact of sex on relative survival and excess mortality following acute myocardial infarction (AMI) using a population-based cohort within a relative survival framework. Patient-level data concerning demographics, co-morbidity, cardiovascular risk factors and treatments at discharge were extracted from the Swedish Web-system for Enhancement and Development of Evidence-based care in Heart disease Evaluated According to Recommended Therapies (SWEDEHEART), a population-based registry of outcomes for patients hospitalized with acute coronary syndrome. Patients were followed-up for their vital status after AMI hospitalisation, with censoring at the end of follow-up on the 31st of December, 2013.

DETAILED DESCRIPTION:
Details of SWEDEHEART and data validation have been described previously. Cases of acute myocardial infarction were defined as STEMI and NSTEMI according to the current European Society of Cardiology, American College of Cardiology and American Heart Association guidelines and determined at local level by the attending Consultant.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they are aged over 18 years who had been hospitalised following acute myocardial infarction between 1st January, 2003 and 31st December, 2013

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years who had been hospitalised following acute myocardial infarction between 1st January, 2003 and 31st December, 2013
Sampling Method: Non-Probability Sample
Enrollment: 180000 (Actual)
Dates: Start 2003-12; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Excess mortality rate ratio | 10 years

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alabas OA, Gale CP, Hall M, Rutherford MJ, Szummer K, Lawesson SS, Alfredsson J, Lindahl B, Jernberg T. Sex Differences in Treatments, Relative Survival, and Excess Mortality Following Acute Myocardial Infarction: National Cohort Study Using the SWEDEHEART Registry. J Am Heart Assoc. 2017 Dec 14;6(12):e007123. doi: 10.1161/JAHA.117.007123. PMID 29242184